CLINICAL TRIAL: NCT00637507
Title: Phase II/Phase III Study of the Effect of Combined High-frequency Oscillation and Tracheal Gas Insufflation on the Survival to Hospital Discharge of Patients With Severe Acute Respiratory Distress Syndrome
Brief Title: Study of a Novel Technique of Mechanical Ventilation in Patients With Severe Acute Respiratory Failure
Acronym: HFO-TGI-2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Athens (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Spyros D. Mentzelopoulos, Assistant Professor of Intensive Care Medicine, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFO-TGI-728-4-10-07
Record Dates: First submitted 2008-03-04; First posted 2008-03-18 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Respiratory Distress Syndrome
Keywords: High-Frequency Ventilation; Tracheal Gas Insufflation; Respiration, Artificial; Respiratory Distress Syndrome; Adult
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration | interventions — High-Frequency Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (No Intervention): Patients treated solely with a pressure- and volume-limited ventilatory strategy (target plateau pressure of 30 cm H2O) aimed at minimizing lung stress and strain, and thus, ventilator-induced lung injury.
- 1 (Experimental): Intermittent application of High-frequency Oscillation (HFO) and Tracheal Gas Insufflation (TGI) according to pre-specified criteria described in the Detailed Description. HFO-TGI sessions are interspersed with lung protective conventional mechanical ventilation until the PaO2/FiO2 ratio stabilizes at >150 mm Hg.
  Interventions: Other: High-frequency Oscillation and Tracheal Gas Insufflation

INTERVENTIONS:
Other: High-frequency Oscillation and Tracheal Gas Insufflation — Patients will receive daily sessions of High-frequency Oscillation and Tracheal Gas Insufflation (HFO-TGI), which will last at least 6 hours. These sessions will comprise a recruitment period of at least 90 min, a stabilization period of at least 4 hours, and a weaning period of at least 60 min. The HFO-TGI strategy will be aimed at initially maximizing PaO2/FiO2 without causing hemodynamic compromise (e.g., >10% reduction in cardiac output/index), and subsequently maintaining PaO2/FiO2 >150 mm Hg, while gradually reducing mPaw to 4-6 cm H2O below its initial setting. The weaning from TGI and HFO will be according to the reversal of the oxygenation criterion that mandated their use (see also Detailed Description).
  Other Names: HFO-TGI
  Arms: 1

SUMMARY:
The investigators have recently demonstrated the beneficial effects of combined high-frequency oscillation (HFO) and tracheal gas insufflation (TGI) on the respiratory physiology [1,2] of patients with severe acute respiratory distress syndrome (ARDS) (NCT00416260). Preliminary short-term survival results were also encouraging. Consequently, in the present clinical trial, the investigators intend to increase the size of the studied population, in order to evaluate the effect of HFO-TGI on survival with adequate statistical power. Furthermore, the investigators intend to elucidate the mechanism of the HFO-TGI-related physiological benefit.

DETAILED DESCRIPTION:
BACKGROUND AND OBJECTIVES

The prognosis of ARDS still remains grave [3-7]. The primary objective of the present study, is to definitively determine the effect of HFO-TGI on the survival of patients with severe ARDS. Consequently, we will increase the size of the studied population (see also NCT00416260), in order to achieve sufficient statistical power. The secondary objective is to test the hypothesis that lung recruitment is the major underlying mechanism for the HFO-TGI-associated improvement in oxygenation [1,2] and respiratory compliance [2].

METHODS

Patients

The protocol has been approved by the Scientific Committees of Evaggelismos Hospital and of Larissa University Hospital. Informed consent will be requested from the next-of-kin of participation-eligible patients. Patients will be informed of the trial and their right to withdraw as soon as clinically feasible. Eligibility criteria are presented in the appropriate section of this report. In brief, the major inclusion criteria will comprise 1) early (diagnosis established within the preceding 72 h) ARDS according to the American-European Consensus Conference Definition [6]; 2) severe oxygenation disturbances {defined as PaO2/FiO2) < 150 mm Hg}, while ventilated with a positive end-expiratory pressure (PEEP) of ≥ 8 cm H2O (criterion for severe ARDS); and 3) age 18-75 years and body weight > 40 kg. Patient monitoring will include electrocardiographic lead II, hemodynamics {continuous intraarterial and central-venous pressure, and cardiac output/index by PICCO-plus (Pulsion Medical Systems, Munich, Germany)}, and peripheral oxygen saturation (SpO2). Deep sedation (propofol/midazolam) [8,9], analgesia (fentanyl/remifentanil) [9], and intermittent neuromuscular blockade (cisatracurium) [8,10] will be used.

CMV Strategy

In the 37-bed intensive care unit (ICU) of Evaggelismos hospital and the 10-bed ICU of Larissa hospital, a pressure-and volume-limited ventilatory strategy is routinely employed. Consequently, before randomization, patients will already be ventilated (Siemens 300C ventilator; or Galileo Gold, Hamilton Medical) with one of the ARDSnet-protocol allowable combinations of FiO2 and PEEP [11]. Administered tidal volumes will be 5.5-7.5 mL•kg-1 predicted body weight, ventilatory rate (e.g., 20-35•min-1) will be adjusted so that pHa is kept in-between 7.20-7.45; the inspiratory to expiratory time ratio will be 1:1 to 1:3; and the target plateau inspiratory pressure will be ≤ 35 cm H2O. Oxygenation goals will be PaO2 = 60-80 mm Hg or SpO2 = 90-95%.

Randomization

Patients will be assigned to the HFO-TGI-group (i.e., the intervention-group) or the Conventional Mechanical Ventilation (CMV)-group (i.e., the control-group) according to a computer-generated, random number-sequence (http://www.randomizer.org). Furthermore, crossover from the CMV)-group to the HFO-TGI-group will be performed whenever requested by the attending physicians. Randomization will be undertaken by the department's statistician and will be supervised by the Independent Main End Point and Safety Monitoring Committee, which will be the same as for NCT00416260, with an additional member at Larissa hospital. Group allocation will be concealed until study entry.

HFO-TGI strategy

Just prior to HFO-TGI initiation, a TGI catheter (internal / external diameter = 1.0 / 2.0 mm, respectively) will be introduced into the endotracheal tube. TGI catheter tip will be placed 0.5-1 cm beyond the endotracheal tube tip. For TGI administration, the proximal end of the TGI catheter will be connected to a variable-orifice O2 flowmeter. The Sensormedics 3100B high-frequency ventilator will be connected to the endotracheal tube. Initial HFO settings will be as follows: 1) FiO2 = 100%, later-on titrated toward the FiO2 of preceding CMV; 2) bias flow = 30-40 L•min-1; 3) oscillation frequency = 4.0-5.0 Hz; 4) oscillatory pressure amplitude = arithmetical PaCO2 value during preceding CMV + 20-30 cm H2O, maximal acceptable value = 95-100 cm H2O [1]; 5) inspiratory to expiratory time ratio = 1:2; and 6) mPaw adjusted to 9-10 cm H2O above preceding CMV mPaw (corresponding to an HFO-mean tracheal pressure of 2-3 cm H2O above the mean tracheal pressure of the preceding CMV). Three-to-five mins after HFO initiation, a recruitment maneuver will be performed by pressurizing the HFO circuit at 40-45 cm H2O for 30-40 secs with oscillator piston off. HFO will then be resumed, and a 3-5 cm H2O endotracheal tube cuff leak will be placed. Immediately thereafter, continuous forward thrust TGI {flow = 50% of the minute ventilation of the preceding CMV [1]} will be superimposed on the HFO. The mPaw control knob will then be adjusted to return mPaw to its originally set value. Fifteen min thereafter, arterial blood gas analysis will be performed and oscillatory pressure amplitude and oscillation frequency will be adjusted, in order to achieve a PaCO2 of < 10-15 mm Hg above the PaCO2 of the preceding CMV and to keep pHa > 7.20. At 90 min after HFO-TGI initiation, physiologic measurements (i.e., blood gas analysis and hemodynamics) will be conducted, and then, mPaw will be gradually reduced (estimated reduction rate: 0-2 cm H2O•h-1) toward 6 cm H2O below its initially set value (corresponding to an HFO-mean tracheal pressure of 2-3 cm H2O below the mean tracheal pressure of the preceding CMV). Subsequently, TGI will be discontinued and standard HFO will be continued for 30 min.

Return to CMV will be considered at the following HFO settings: mPaw = 3-4 cm H2O above preceding CMV mPaw (corresponding to an HFO-mean tracheal pressure of 2-3 cm H2O below the mean tracheal pressure of the preceding CMV); and TGI = 0 L•min-1. Return to HFO-TGI will be considered necessary if after 12 h of CMV, PaO2/FiO2 is < 150 mm Hg at a PEEP of ≥ 8 cm H2O. In the HFO-TGI-group, patients will receive repeated daily sessions of HFO-TGI until they no longer satisfy the severe ARDS criterion during CMV for at least 48 h. Predicted minimum duration of HFO-TGI sessions is 6 h. During HFO-TGI sessions, physiologic measurements will be performed every 1.5-4 h, and their average values will be used in the subsequent statistical analysis. For HFO-TGI-group members, total HFO-TGI duration will have to be > 12 h.

Recruitment Maneuvers

Recruitment maneuvers (with continuous positive airway pressure of 40-45 cm H2O and a duration of 40 secs) will be performed as follows:

In the HFO-TGI group, recruitment maneuvers will be performed at the onset and at 3 and 5 h following the onset of each HFO-TGI session, and just after to return to CMV. In the CMV-group, ≥ 4 recruitment maneuvers (one every 4-6 h; starting at 07:00) will be performed daily. In both groups, recruitment maneuvers will be continued for the first 4 days post-randomization [12].

Weaning from CMV

Weaning from CMV will be by pressure-supported ventilation when a PaO2 of > 60 mm Hg can be maintained at an FiO2 of ≤ 50% and a PEEP of ≤ 8 cm H2O.

Data Collection

Data on demographic, physiologic, and radiographic characteristics, coexisting conditions, and medication will be recorded within 4 h prior to randomization. For the first 10 days post-randomization, at least 3 sets physiologic measurements (blood-gas analysis, hemodynamics, and respiratory mechanics during CMV) will be obtained daily. Laboratory, radiographic/imaging, and physiologic data will be collected daily until ICU discharge or death. Patients will be monitored daily for signs of failure of nonpulmonary organs and systems. Patient clinical course will be documented until hospital discharge or death.

Follow-up of Lung Recruitment with CT of the Thorax

During the intervention period of the present study, we intend to assess and monitor the evolution of lung recruitment, as recently suggested and described in detail by Gattinoni and colleagues [13]. The recruitment-assessment protocol will be as follows: 1) HFO-TGI-group: CT of the thorax at baseline, and at days 5 and 8 post-randomization; 2) CMV-group: CT of the thorax at baseline, and at day 8 post-randomization. Patients will be considered as eligible for CT-evaluation if PaO2/FiO2 is in-between 100-150 mmHg, and if there is no additional concern with respect to patient transportation safety to the CT suite, as confirmed by the attending physicians on a case-by-case basis. The rationale for this investigational intervention comprises the elucidation of the mechanism of the HFO-TGI-induced physiological benefit.

Outcome measures are mentioned in the appropriate section.

In concordance with a suggestion of a recent Editorial (Intensive Care Med (2014) 40:743-745), the Original and (its revision to) the Final Form of the Study Protocol (also corresponding to NCT00416260 which was registered as the first study period) detailing the Pre-specified Study Planning (which explains the reason for any prior changes in the current registration data) can be found by scrolling down to the end of the following webpage: http://www.evaggelismos-hosp.gr/index.php/istoriko-eepne

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Body weight > 40 kg
* Endotracheal intubation and mechanical ventilation
* Diagnosis of ARDS established within preceding 72 h
* Severe oxygenation disturbances: PaO2/FiO2 <150 mm Hg sustained for 12 h, despite being ventilated with PEEP ≥8 cm H2O

Exclusion Criteria:

* Active air leak or recent severe air leak (severe air leak: > 1 chest tube per hemithorax with persistent gas leak for > 72 h)
* Severe hemodynamic instability (i.e., systolic arterial pressure < 90 mm Hg despite volume loading and norepinephrine infusion at ≥ 0.5 μg/kg/min)
* Significant heart disease (i.e., ejection fraction <40 %, and/or history of pulmonary edema, and/or active coronary ischemia or myocardial infarction)
* Significant chronic obstructive pulmonary disease (COPD) or asthma {i.e., previous admissions for COPD/asthma, chronic corticosteroid therapy for COPD/asthma, and documented chronic CO2 retention leading to a baseline PaCO2 of > 50 mm Hg (for COPD)}
* Uncontrollable intracranial hypertension (i.e., intracranial pressure >20 mm Hg despite deep sedation, analgesia, hyperosmolar therapy, and minute ventilation titrated to PaCO2 = 35 mm Hg)
* Chronic Interstitial Lung Disease associated with bilateral pulmonary infiltrates
* Lung biopsy or resection on current admission
* Immunosuppression caused by

  * neutropenia [i.e., polymorphonuclear leukocyte count < 1,000/μL (1 x 1012/L)] after chemotherapy or bone marrow transplantation for hematologic cancers
  * corticosteroid or cytotoxic therapy for a nonmalignant disease
  * the acquired immunodeficiency syndrome
* Inability to wean from prone positioning or inhaled nitric oxide
* Pregnancy or morbid obesity (body mass index >40 kg/m2)
* Enrollment in another interventional study
* Crossover from the CMV-group to the HFO-TGI-group at > 72 h after the onset of the severe oxygenation disturbances

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Survival to days 28 and 60 post-randomization, and to Hospital Discharge | 28 days to more than 60 days post-randomization

SECONDARY OUTCOMES:
Lung recruitment during the study-intervention period | 8 days post-randomization
Evolution of Gas-exchange, Hemodynamics, and Respiratory Mechanics during the Study Intervention Period | 8-10 days post-randomization
Ventilator Free Days | 60 days post-randomization
Organ or System Failure Free Days | 60 days post-randomization
Occurrence of barotrauma (i.e., any new pneumothorax, pneumomediastinum, or subcutaneous emphysema, or pneumatocele > 2 cm) | 60 days post-randomization
Occurence of Tracheal Mucosal Injury due to use of Tracheal Gas Insufflation | 8-10 days post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Spyros D Mentzelopoulos, MD, PhD, Principal Investigator — University of Athens Medical School, Athens, Greece; Sotiris Malachias, MD, Principal Investigator — Department of Intensive Care Medicine, Evaggelismos Hospital, Athens, Greece; Spyros G Zakynthinos, MD, PhD, Study Director — University of Athens Medical School, Athens, Greece; Charis Roussos, MD, PhD, Study Chair — University of Athens Medical School, Athens, Greece
Locations (2):
- Greece (2):
  - Department of Intensive Care Medicine, Evaggelismos Hospital, Athens, Attica
  - University General Hospital of Larissa, Larissa, Thessaly

REFERENCES:
- [Background] Mentzelopoulos SD, Roussos C, Koutsoukou A, Sourlas S, Malachias S, Lachana A, Zakynthinos SG. Acute effects of combined high-frequency oscillation and tracheal gas insufflation in severe acute respiratory distress syndrome. Crit Care Med. 2007 Jun;35(6):1500-8. doi: 10.1097/01.CCM.0000265738.80832.BE. PMID 17440419
- [Background] Brun-Buisson C, Minelli C, Bertolini G, Brazzi L, Pimentel J, Lewandowski K, Bion J, Romand JA, Villar J, Thorsteinsson A, Damas P, Armaganidis A, Lemaire F; ALIVE Study Group. Epidemiology and outcome of acute lung injury in European intensive care units. Results from the ALIVE study. Intensive Care Med. 2004 Jan;30(1):51-61. doi: 10.1007/s00134-003-2022-6. Epub 2003 Oct 16. PMID 14569423
- [Background] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Background] Gattinoni L, Tognoni G, Pesenti A, Taccone P, Mascheroni D, Labarta V, Malacrida R, Di Giulio P, Fumagalli R, Pelosi P, Brazzi L, Latini R; Prone-Supine Study Group. Effect of prone positioning on the survival of patients with acute respiratory failure. N Engl J Med. 2001 Aug 23;345(8):568-73. doi: 10.1056/NEJMoa010043. PMID 11529210
- [Background] Bernard GR, Artigas A, Brigham KL, Carlet J, Falke K, Hudson L, Lamy M, Legall JR, Morris A, Spragg R. The American-European Consensus Conference on ARDS. Definitions, mechanisms, relevant outcomes, and clinical trial coordination. Am J Respir Crit Care Med. 1994 Mar;149(3 Pt 1):818-24. doi: 10.1164/ajrccm.149.3.7509706.
- [Background] Mancebo J, Fernandez R, Blanch L, Rialp G, Gordo F, Ferrer M, Rodriguez F, Garro P, Ricart P, Vallverdu I, Gich I, Castano J, Saura P, Dominguez G, Bonet A, Albert RK. A multicenter trial of prolonged prone ventilation in severe acute respiratory distress syndrome. Am J Respir Crit Care Med. 2006 Jun 1;173(11):1233-9. doi: 10.1164/rccm.200503-353OC. Epub 2006 Mar 23. PMID 16556697
- [Background] Fessler HE, Derdak S, Ferguson ND, Hager DN, Kacmarek RM, Thompson BT, Brower RG. A protocol for high-frequency oscillatory ventilation in adults: results from a roundtable discussion. Crit Care Med. 2007 Jul;35(7):1649-54. doi: 10.1097/01.CCM.0000269026.40739.2E. PMID 17522576
- [Background] Jacobi J, Fraser GL, Coursin DB, Riker RR, Fontaine D, Wittbrodt ET, Chalfin DB, Masica MF, Bjerke HS, Coplin WM, Crippen DW, Fuchs BD, Kelleher RM, Marik PE, Nasraway SA Jr, Murray MJ, Peruzzi WT, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists (ASHP), American College of Chest Physicians. Clinical practice guidelines for the sustained use of sedatives and analgesics in the critically ill adult. Crit Care Med. 2002 Jan;30(1):119-41. doi: 10.1097/00003246-200201000-00020. No abstract available. PMID 11902253
- [Background] Murray MJ, Cowen J, DeBlock H, Erstad B, Gray AW Jr, Tescher AN, McGee WT, Prielipp RC, Susla G, Jacobi J, Nasraway SA Jr, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists, American College of Chest Physicians. Clinical practice guidelines for sustained neuromuscular blockade in the adult critically ill patient. Crit Care Med. 2002 Jan;30(1):142-56. doi: 10.1097/00003246-200201000-00021. No abstract available. PMID 11902255
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Gattinoni L, Caironi P, Cressoni M, Chiumello D, Ranieri VM, Quintel M, Russo S, Patroniti N, Cornejo R, Bugedo G. Lung recruitment in patients with the acute respiratory distress syndrome. N Engl J Med. 2006 Apr 27;354(17):1775-86. doi: 10.1056/NEJMoa052052. PMID 16641394
- [Background] Grasso S, Mascia L, Del Turco M, Malacarne P, Giunta F, Brochard L, Slutsky AS, Marco Ranieri V. Effects of recruiting maneuvers in patients with acute respiratory distress syndrome ventilated with protective ventilatory strategy. Anesthesiology. 2002 Apr;96(4):795-802. doi: 10.1097/00000542-200204000-00005. PMID 11964585
- [Background] Peto R, Pike MC, Armitage P, Breslow NE, Cox DR, Howard SV, Mantel N, McPherson K, Peto J, Smith PG. Design and analysis of randomized clinical trials requiring prolonged observation of each patient. I. Introduction and design. Br J Cancer. 1976 Dec;34(6):585-612. doi: 10.1038/bjc.1976.220. PMID 795448
- [Background] Geller NL, Pocock SJ. Interim analyses in randomized clinical trials: ramifications and guidelines for practitioners. Biometrics. 1987 Mar;43(1):213-23. PMID 3567306
- [Background] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Result] Mentzelopoulos SD, Malachias S, Tzoufi M, Markaki V, Zervakis D, Pitaridis M, Zakynthinos S. High frequency oscillation and tracheal gas insufflation for severe acute respiratory distress syndrome [abstract]. Intensive Care Med 2007;33(Suppl 2):S142
- [Derived] Mentzelopoulos SD, Malachias S, Zintzaras E, Kokkoris S, Zakynthinos E, Makris D, Magira E, Markaki V, Roussos C, Zakynthinos SG. Intermittent recruitment with high-frequency oscillation/tracheal gas insufflation in acute respiratory distress syndrome. Eur Respir J. 2012 Mar;39(3):635-47. doi: 10.1183/09031936.00158810. Epub 2011 Sep 1. PMID 21885390